CLINICAL TRIAL: NCT00459797
Title: Comparison of Conventional GlideScope to Single-Use GlideScope Cobalt for Orotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Philip Jones, LHSC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-07-040; 13025
Record Dates: First submitted 2007-04-12; First posted 2007-04-13 (Estimated); Last update posted 2009-04-21 (Estimated); Status verified 2009-04

CONDITIONS: Healthy
Keywords: GlideScope; cobalt; single-use; intubation; airway; Elective surgical patients requiring orotracheal intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Glidescope (Active Comparator)
  Interventions: Device: Conventional (reusable) Glidescope
- Single-use Glidescope (Experimental)
  Interventions: Device: Single-use Glidescope videolaryngoscope

INTERVENTIONS:
Device: Conventional (reusable) Glidescope
  Arms: Conventional Glidescope
Device: Single-use Glidescope videolaryngoscope
  Arms: Single-use Glidescope

SUMMARY:
Patients presenting for elective surgery requiring orotracheal intubation will be randomized to being intubated with either the conventional (reusable) GlideScope videolaryngoscope or the single-use GlideScope videolaryngoscope. The primary outcome is time to intubation.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who is ≥ 18 yrs. coming for elective surgery.
* Endotracheal tube is indicated for the procedure in the opinion of the attending anesthesiologist.
* Any operator who has performed ≥ 10 GlideScope intubations.

Exclusion Criteria:

* Any patient in whom the use of the GlideScope is contraindicated in the opinion of the attending anesthesiologist.
* Any patient with cervical spine abnormalities.
* Any patients with known or probable difficult airways (this rare occurrence is unlikely to be evenly distributed between the groups and could skew the data).
* Any patient requiring rapid sequence induction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Time to intubation (seconds) | Immediate

SECONDARY OUTCOMES:
Ease of intubation | after intubation
Number of intubation attempts per group | after intubation
Incidence of trauma in each group | after intubation
Number of failures to intubate per group | after intubation
Use of external laryngeal pressure per group | after intubation
Laryngoscopic grade distribution in each group | after intubation

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Jones, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Jones PM, Turkstra TP, Armstrong KP, Armstrong PM, Harle CC. Comparison of a single-use GlideScope Cobalt videolaryngoscope with a conventional GlideScope for orotracheal intubation. Can J Anaesth. 2010 Jan;57(1):18-23. doi: 10.1007/s12630-009-9204-9. Epub 2009 Oct 31. PMID 19882199